CLINICAL TRIAL: NCT05023096
Title: Effects of Electronic Nicotine Delivery System Flavor Regulations on Tobacco Behavior, Toxicity, and Abuse Liability Among African American Menthol Smokers
Brief Title: Potential Effects of Electronic Nicotine Delivery System Flavor Regulations on African American Menthol Smokers
Acronym: RVA Flavors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20022060; 1R01DA050996-01A1 (NIH)
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Electronic Nicotine Delivery System Flavors
Keywords: Electronic Nicotine Delivery System; Electronic Cigarette; Flavor; Abuse Liability; Toxicant Exposure; Tobacco; African American; Menthol
MeSH Terms: conditions — Vaping | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Menthol+Tobacco (Active Comparator): Menthol+Tobacco - where both menthol and tobacco flavored liquids for electronic nicotine delivery systems are available to choose from
  Interventions: Other: Tobacco product administration and assessment
- Tobacco (Experimental): Tobacco - where only tobacco flavored liquid is available for electronic nicotine delivery systems
  Interventions: Other: Tobacco product administration and assessment
- Unflavored (Experimental): Unflavored - where only unflavored liquid is available for electronic nicotine delivery systems
  Interventions: Other: Tobacco product administration and assessment

INTERVENTIONS:
Other: Tobacco product administration and assessment — Participants are first instructed to smoke their usual brand of menthol cigarettes normally for the next 7 days and avoid using any other tobacco products. After this baseline week, participants are randomized to 1 of 3 ENDS flavor conditions, all contain 5% nicotine (Mentol+Tobacco, Tobacco, Unflavored) with equal probability and provided with a supply of their condition specific ENDS and asked to use it in place of their usual menthol cigarettes for the next 6 weeks.

SUMMARY:
This study aims to better understand how the availability of electronic nicotine delivery system (aka electronic cigarettes) flavors (e.g., menthol, tobacco) impacts tobacco use behaviors, toxicant exposure, and abuse liability among African American menthol smokers.

DETAILED DESCRIPTION:
Black/African American (AA) menthol smokers are disproportionately harmed by tobacco products and could experience significant health benefits from increased availability of well-regulated electronic nicotine delivery systems (ENDS). The current study will evaluate whether ENDS flavor availability affects measures of tobacco use, biomarkers of cigarette/ENDS exposure, and addiction among AA menthol smokers by performing a 3-arm, 6-week clinical trial of ENDS provision with follow-up to 30 days. Results of this work will help FDA make predictions about the impact of moving from the current regulatory market were menthol/tobacco flavored ENDS cartridges are available, to one where only tobacco or unflavored cartridges are available, in order to maximize health-promoting effects and minimize unintended consequences among AA menthol smokers.

ELIGIBILITY:
Inclusion Criteria:

* 21+ years of age
* identify as Black/African American (single or multi-race)
* have used ≥5 cigarettes per day for ≥1 year
* biochemically confirmed cigarette smoking status
* regular cigarette brand is flavored to taste like menthol or mint
* ENDS use in the past 3 months
* report no intent to quit smoking in the next 6 months
* previous quit attempt using evidence-based method
* have a working mobile phone with a texting/data plan
* are willing receive phone calls/text messages and complete internet-based/online surveys related to the study.
* read and write in English

Exclusion Criteria:

* are unwilling to use ENDS as part of the trial
* unstable or significant medical condition in the past 12 months
* report any other illegal drug use in past 30 days
* report intent to become pregnant or current pregnancy/breastfeeding
* report any other condition that may affect participant safety or not allow them to fully participate in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Average Daily Cigarette Use | Week 1 vs. Week 6
  Number of cigarettes used in the past day, collected via daily text survey, averaged over the past week
Change in Carbon Monoxide Exposure | Week 1 vs. Week 6
  A biomarker of combusted cigarette use collected from exhaled breath
Willingness to Substitute from Cigarettes to ENDS | Week 6
  Measure of substitution for condition-specific tobacco products will be assessed using drug purchase tasks. Choices made during this task are not reinforced.

SECONDARY OUTCOMES:
Change in Average Daily ENDS Use | Week 1 vs. Week 6
  Number of ENDS puffs in the past day, collected via daily text survey, averaged over the past week
Change in NNAL Exposure | Week 1 vs. Week 6
  A biomarker of combusted cigarette use collected from urine
Change in Proplyne Glycol Exposure | Week 1 vs. Week 6
  A biomarker of ENDS use collected from urine
Willingness to Pay for ENDS | Week 6
  Willingness to pay for condition-specific tobacco products will be assessed using drug purchase tasks. Choices made during this task are not reinforced.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Barnes, PhD, Principal Investigator — Virginia Commonwealth University; Caroline O Cobb, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States